CLINICAL TRIAL: NCT04826419
Title: Non-invazive Ozone Therapy and Digital Ulcer in Patients With SSc
Brief Title: Effect of Ozone Therapy for the Treatment of Digital Ulcer in Patients With SSc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hakan Alkan, Clinical Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pamukkale U
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: randomised-controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invazive ozone therapy in a group (Active Comparator): ozone therapy
  Interventions: Other: ozone therapy
- Control group (No Intervention): control groups do not take ozone therapy

INTERVENTIONS:
Other: ozone therapy — The treatment session of oxygen-ozone was 80 mg/mL ozone (total volume: 60-100 mL) in a special bag using the ozone generator device (Humazon Promedic, German) five times a week for the first week.The treatment session of oxygen-ozone was 40 mg/mL ozone (total volume: 60-100 mL) in a special bag using the ozone generator device (Humazon Promedic, German) twice a week after first week.
  Arms: Non-invazive ozone therapy in a group

SUMMARY:
Functionality in patients with SSc? Systemic Sclerosis (SSc) is a chronic connective tissue disease characterized by microvascular involvement, immunological dysfunction, extracellular matrix deposition in the skin and internal organ involvement. Vascular disease has an important role in the pathogenesis of SSc. Especially as a result of involvement of micro-vessel and digital arteries, digital ulcer (DU) formation may be seen. DUs are responsible for pain, poor quality of life, impairment of life activities and morbidity in patients with SSc. , they are correlated to disease severity and outcome. Approximately half of SSc patients have DU during the course of the disease. Recurrent DU is observed in 10% of the patients. In 75% of these patients, DU occurs 5 years after diagnosis. Patients with anti-SCL 70+ develop DU 5 years earlier than those with anti-centromere positive. The development of DU may take a long time to heal if there is underlying calcinosis. In a study, it was seen that the recovery of DU was 93.6 days if there is underlying calcinosis, and 76.2 days if not. DUs can be infected and thus complicated by osteomyelitis. In a retrospective study, it was reported that 42% of infected DUs were associated with osteomyelitis. DU management is a great challenge for the clinician and requires a multidisciplinary approach. Ozone has a place in medical use since the 19th century, as it is an oxidant and disinfectant. In recent studies, it has been reported to be antiviral and bactericidal. Therefore, it has indications such as coronary artery disease, chronic hepatitis and chronic low back pain. It has also been shown to have a positive role in trophic ulcer, ischemic ulcer and diabetic ulcer healing. The mechanism by which ozone therapy provides wound healing is not fully understood. In addition, it improves microcirculation in the capillary vessels by improving flexibility and stability of the cell membrane and limiting the aggregation and adhesion of platelets.

In the literature, it was stated in a study that ozone therapy was effective for the treatment of DU in SSc patients. In our study, we aimed to investigate the effect of ozone therapy on patients who are resistant to medical treatment and who have impaired quality of life for a long time.

DETAILED DESCRIPTION:
Material-Method 34 SSc patients who were followed up in Pamukkale University Rheumatology due to DU are going to be included in the study. SSc is diagnosed and based on the American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) Criteria for the classification of SSc. Skin thickness will be evaluated with the Modified Rodnan Score.

DUs will be graded according to a scale developed by Amanzi et al. In 2010. Written informed consents were obtained from all patients before entry into the study, according to the Declaration of Helsinki and guidelines of the local ethics committee. The study was approved by Pamukkale University ethics committee. Among the patients included in the study, those with gangrenous ulcers, calcinosis-free ulcers, traumatic ulcers, vasculitis, active osteomyelitis, hyperthyroidism, pregnancy, and allergies to ozone therapy will be excluded from the study.

Baseline evaluation The demographic profile of SSc patients, therapy, scleroderma type, the onset of reynoud phenomenon (RF) RF disease duration, RFI time with the number of daily attacks, active and inactive digital ulcers count, ulcer size, pain, number of pitting, laboratory findings, and functional scales will recorded. Antinuclear antibodies (ANA), anti-centromere antibodies (ACA) and anti-topoisomerase antibodies (Scl70) will be studied from laboratory findings. An indirect immunofluorescent assay, for semi quantitative determination of anti-nuclear IgG antibodies (ANA) in patients' serum NOVA LITE™ IFA HEp-2 ANA Complete Kit was used. Antibodies to extractable nuclear antigens ACA and Scl70 are going to be determined by a commercial clinical enzyme linked immunosorbent assay (ELISA).

Functional parameters such as health assessment questionnaire (HAQ), visual analogue scale (VAS) and Modified Hand Mobility in Scleroderma Test (HAMISm) will be evaluated before treatment and on the 30th day.

Interventıon Group The treatment or clinical status of the SSc patients followed up with DU was reached by a blinded health professional by phone. Those who wanted to participate actively in the study formed the ozone group, but those who did not want to participate due to the pandemic constituted the control group.

Ozone Group The treatment session of oxygen-ozone was 80 mg/mL ozone (total volume: 60-100 mL) in a special bag using the ozone generator device (Humazon Promedic, German).

Treatment group Similar demographic results and treatment protocols area with treatment group consisted of SSc patients.

Outcomes Primary outcomes Ulcer healing was our primary outcome, which was assessed depending on Zhang andcolleagues ulcers grading where they graded ulcers into four levels, Grade 0 (no change), Grade 1 (wound size decreased less than ½); Grade 2 (wound size decreased more than ½) and Grade 3 (wound healing) (31). Ozone treatment were considered efficient if patients reached grade 1 to 3.

Secondary outcomes For our secondary outcomes both group were subjected to the following after two weeks and four weeks of intervention: they were reassessed for number of Raynaud's attacks/day, duration of Raynaud's attack, ulcer size in mm, ulcer pain was assessed by VAS and functional status evaluated by HAQ and HAMISm.

ELIGIBILITY:
Inclusion Criteria:

• SSc patients who have no comorbidity

Exclusion Criteria:

* gangrenous ulcers
* calcinosis-free ulcers
* traumatic ulcers
* vasculitis
* active osteomyelitis
* hyperthyroidism
* pregnancy
* allergies to ozone therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Ulcer healing | one month
  Ulcer healing was our primary outcome, which was assessed depending on Zhang andcolleagues ulcers grading where they graded ulcers into four levels, Grade 0 (no change), Grade 1 (wound size decreased less than ½); Grade 2 (wound size decreased more than ½

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Kaymaz, M.D, Principal Investigator — Pamukkale U
Locations (1):
- Pamukkale Unıversity, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no plan

REFERENCES:
- [Background] Zhang J, Guan M, Xie C, Luo X, Zhang Q, Xue Y. Increased growth factors play a role in wound healing promoted by noninvasive oxygen-ozone therapy in diabetic patients with foot ulcers. Oxid Med Cell Longev. 2014;2014:273475. doi: 10.1155/2014/273475. Epub 2014 Jun 24. PMID 25089169